CLINICAL TRIAL: NCT00287014
Title: Late Outcomes of Rift Valley Fever in Kenya: Ijara Clinical Survey
Brief Title: Rift Valley Fever in Kenya
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0042
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-10

CONDITIONS: Rift Valley Fever
Keywords: Rift valley fever, Kenya
MeSH Terms: conditions — Rift Valley Fever

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to find out how, why, and when Rift Valley Fever (RVF) spreads. Participants will be 250 adults and children, aged 1 year and older, from the Ijara District, Kenya. They will be given a questionnaire, undergo a medical examination that includes an eye exam, and have a 1-teaspoon sample of blood taken from a vein. Participation will take about 3 hours.

DETAILED DESCRIPTION:
The objective of this research is to better define the extent and timing of Rift Valley Fever (RVF) virus transmission and its related chronic disease/infection attack rate, during an interepidemic period in a high-risk region that has seen repeated RVF outbreaks. The results will be used to develop and refine predictive algorithms for RVF Virus transmission, based on epidemiological, environmental, and remote sensing data, with the ultimate goal of providing improved early detection of significant RVF outbreaks. It is expected that the analysis of test-performance characteristics will determine the best use of serologic assays in Kenya's next RVF epizootic/epidemic. The primary outcome measure will be the current RVF-specific seropositivity profile for a cross-sectional survey population in Ijara District in northeast Kenya. The secondary outcome measures to be studied will be: 1) an assessment of the behavioral factors associated with risk of seropositivity (previous infection) in the study population; and 2) the association of selected long-term ophthalmological and clinical outcomes with seropositivity. The study design for this protocol involves questionnaire administration to consenting participants of Ijara District, followed by performance of medical exams, ophthalmologic exams, and phlebotomy on all participants. ELISA testing for RVF will then be performed on the blood samples obtained, and all ELISA screen-positive samples will have confirmatory testing by plaque-reduction neutralizing antibody testing.

ELIGIBILITY:
Inclusion Criteria:

Those adults and children residing in selected survey households in the area of Ijara Town and its 5 km environs who are 1 year of age and older will be eligible, provided:

1. Informed consent is obtained and signed, and assent form is obtained and signed from children age 7 and older,
2. Subject has understanding of study procedures, and
3. Subject is able to comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Age less than 1 year.
2. Subjects who immigrated to the study area less than 2 years previously.
3. Acutely ill Ijara residents.
4. Adults and children who cannot provide informed consent or who cannot participate fully in the study procedures will also be excluded.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 2006-03; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Locations (1):
- Ijara District, Ijara, Kenya